CLINICAL TRIAL: NCT06992089
Title: Pacemaker Implantation in Patients With Heart Failure With Preserved Ejection Fraction, Chronotropic Incompetence and Small Ventricular Volume. The SHOP-HF Trial
Brief Title: SHort Of Pace - Heart Failure (SHOP-HF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SHOP-HF
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacing on (Experimental): Pacemarker stimulation programmed as AAIR / DDDR / VVIR with the basic stimulation frequency and the rate response as follows (pacing on):
  * Basic heart rate: derived from the averaged resting heart rates of healthy adults according to height and LVEF.
  * Rate response through a combination of minute ventilation and accelerometer: with a response factor of 3 and a medium-low activity threshold.
  Interventions: Device: Dual-chamber cardiac pacemaker (Essentio MRI L111 Boston Scientific®), Single-chamber cardiac pacemaker (Essentio MRI L110 Boston Scientific®)
- Pacing off (Placebo Comparator): VVI 30 bpm
  Interventions: Device: Dual-chamber cardiac pacemaker (Essentio MRI L111 Boston Scientific®), Single-chamber cardiac pacemaker (Essentio MRI L110 Boston Scientific®)

INTERVENTIONS:
Device: Dual-chamber cardiac pacemaker (Essentio MRI L111 Boston Scientific®), Single-chamber cardiac pacemaker (Essentio MRI L110 Boston Scientific®) — Dual-chamber cardiac pacemaker (Essentio MRI L111 Boston Scientific®), with rate-adaptive pacing of the right atrium. There will be an associated right atrial lead (INGEVITY™ MRI Pacing Lead Boston®) and right ventricular lead (INGEVITY™ MRI Pacing Lead Boston®).
  Single-chamber cardiac pacemaker (Essentio MRI L110 Boston Scientific®), with rate-adaptive pacing of the ventricles. There will be a right ventricular lead (INGEVITY™ MRI P Boston®).

SUMMARY:
This study is designed as a multicenter, prospective, controlled, randomized, two-arms, cross-over, two parallel cohorts, efficacy Clinical research with CE-marked medical device . The crossover trial will be performed in a blind fashion, so each participant will be evaluated during both blinded pacing-on and pacing-off phases, each of which will last 3 months. The population includes patients with the diagnosis of stable HFpEF according to criteria of the European Society of Cardiology and New York Heart Association (NYHA) functional class II-III/IV, left ventricular hypertrophy with small ventricular volume, sinus rhythm with low basal heart rate and chronotropic incompetence (CI).

All patients will undergo pacemaker implantation, and computer-generated randomization sequence previously designed will be used to allocate participants (in a 1:1 ratio) to receive: (a) programming of the pacemaker with pacing On followed by pacing Off in two periods of 3 months; or (b) programming of the pacemaker with pacing Off followed by pacing On in two periods of 3 months. The study will be conducted in three centers in Spain. Discounting the time due to staggered entry, the total duration of a patient's follow-up will be 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Stable symptomatic heart failure (NYHA functional class ≥II) during the last month.
* Diagnosis criteria of HFpEF according to ESC guidelines:

  1. symptoms and signs of HF.
  2. left ventricular ejection fraction ≥50% by Simpson method.
  3. proBNP >125 pg/mL in the last month.
  4. at least one additional criterion: 1. relevant structural heart disease (left ventricular hypertrophy and/or left atrial enlargement); and/or 2. Diastolic dysfunction.
* Left ventricular hypertrophy was defined as wall thickness > 10 mm.
* Small ventricular volume was defined as indexed left ventricular end diastolic volume < 45 ml/m2.
* Adults ≥18 years old.
* Previous admission for acute heart failure.
* Chronotropic incompetence assessed by CPET, defined as: [(HRmax - HRrest)]/[(220 - age) - (HRrest)] < 0.62.
* Resting heart rate < 65 bpm in sinus rhythm or 70 bmp in atrial fibrillation.

Exclusion Criteria:

* Inability to perform a valid baseline exercise test.
* Significant primary pulmonary disease; including pulmonary arterial hypertension, chronic thromboembolic pulmonary disease or chronic obstructive pulmonary disease.
* Patient with prior history of left ventricular ejection fraction <50%.
* History of an acute coronary syndrome in the previous 12 months.
* Effort angina or signs of ischemia during CPET.
* RER threshold at <1.05 at the CPET.
* Significant primary moderate to severe valvular disease.
* Any other comorbidity with a life expectancy lower than 1 year.
* Heart rate at rest > 75 lpm.
* Other pacemaker indication.
* Pregnant women.
* Baseline rhythm different from sinus rhythm or atrial fibrillation.
* Active treatment with beta-blockers, digitalis or non dihidropiridine calcium channel blockers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | 3 months after the pacemarker stimulation
  The primary endpoint of the study is absolute and relative changes in peak oxygen uptake (peakVO2) after three months of pacemaker stimulation.

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | From randomization until the end of study in month 7
  Absolute changes in quality of live assessed by Minnesota Living with Heart Failure Questionnaire (MLHFQ)
E/E' ratio | From baseline until the end of study in month 7
  Absolute changes in echocardiogram parameters (E/E' ratio)
Left ventricular volume index | From baseline until the end of study in month 7
  Absolute changes in echocardiogram parameters (Left ventricular volume index)
Left atrial volume index | From baseline until the end of study in month 7
  Absolute changes in echocardiogram parameters (Left atrial volume index)
Pro-B-type natriuretic peptide | From baseline until the end of study in month 7
  Absolute and relative changes in prognostic biomarkers (pro-B-type natriuretic peptide)
Serum carbohydrate antigen 125 | From baseline until the end of study in month 7
  Absolute and relative changes in prognostic biomarkers (serum carbohydrate antigen 125).

OTHER OUTCOMES:
Acute HF hospitalizations | From baseline until the end of study in month 7
  Total number of episodes of acute HF hospitalizations.
Worsening HF not requiring hospitalization | From baseline until the end of study in month 7
  Total episodes of worsening HF not requiring hospitalization
Mortality | From baseline until the end of study in month 7
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Julio Núñez, Doctor, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico de la Comunidad Valenciana, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No